CLINICAL TRIAL: NCT06151418
Title: Novel Hormonal Therapy (NHT) for Treating Patients With Metastatic Castration-Sensitive Prostate Cancer (mCSPC): An Analysis of National Veterans Affairs Health Care Network Data
Brief Title: A Study to Learn About Novel Hormonal Therapies (NHTs) for Metastatic Castration-sensitive Prostate Cancer (mCSPC) in People Who Were in the Armed Forces
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C3431052; NCT06151418 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Prostatic Neoplasms
Keywords: metastatic castration-sensitive prostate cancer; mCSPC; metastatic hormone-sensitive prostate cancer; mHSPC; enzalutamide; abiraterone; treatment duration; time to next therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novel hormonal therapy cohort: Patients initiating novel hormonal therapy (abiraterone, apalutamide or enzalutamide) for mCSPC
  Interventions: Drug: Novel hormonal therapy

INTERVENTIONS:
Drug: Novel hormonal therapy — As provided in real-world setting
  Other Names: Abiraterone(Yonsa, Zytiga); Apalutamide(Erleada); Enzalutamide(Xtandi)

SUMMARY:
The purpose of this study is to learn about- for how long are NHTs taken by men to treat mCSPC. NHTs in this study include study medicines:

* abiraterone,
* apalutamide,
* enzalutamide.

Prostate cancer is one of the most common cancers in men. The prostate is a gland in the male body that helps make semen. Metastatic cancer is a cancer that has spread to other parts of the body. Most prostate cancers need male hormones to grow. When cancer cells respond to treatment that lowers male hormones, this is known as castration-sensitive prostate cancer.

This is a real-world study, not a clinical trial. This means that researchers will look at what happens when men receive the treatments prescribed by their own doctor as part of their usual healthcare treatment. In this study, researchers will use information from National Veteran's Affairs (VA) Health Care Network.

The study will include patients' information from the database for men who:

* were identified to have mCSPC.
* started treatment with NHT for mCSPC.
* were 18 years of age or older at start of NHT.

Men in this study will be taking NHT for treatment of their mCSPC. The study will explain:

* how long men take the therapy.
* how long it takes to start next therapy.

This study will use patient information about medications and treatments from VA data. This study will use information one year before start of NHT until information is available.

ELIGIBILITY:
Inclusion Criteria:

* Male with ≥ 1 diagnosis claim for prostate cancer
* Had documented secondary metastasis code on or after the initial prostate cancer diagnosis
* Had initiated novel hormonal therapy (abiraterone, apalutamide, or enzalutamide) within 90 days prior to the metastasis date or on or after the metastasis date. The initiation date of the earliest novel hormonal therapy will be defined as the index date
* ≥18 years old on index date
* Continuous enrollment for at least 365 days before index date
* Evidence to be castration-sensitive:

  * No prior surgical castration any time prior to the index date or no medical castration with ≥8 weeks of continuous use within -90 to -365 days prior to the index date, OR
  * Diagnosis of hormone sensitive malignancy status within 90 days before the index date

Exclusion Criteria:

* Evidence of castration-resistance prior to the index date

  * Received other prostate cancer treatment including NHT, non-steroidal anti-androgen (NSAA), chemotherapy, immunotherapy, radium 223, lutetium Lu 177 vipivotide tetraxetan, ketoconazole, or PARP inhibitor prior to the index date
  * Had diagnosis code indicating hormone resistance prior to the index date
  * A rise in prostate-specific antigen from the nadir by ≥2 ng/mL after castration
* Had a prior history of other cancers (except non-melanoma skin cancer)
* Participation in a clinical trial during the 30 days before the index date

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men with metastatic castration-sensitive prostate cancer who initiated novel hormonal therapy (abiraterone, apalutamide, or enzalutamide) and met eligibility criteria will be included in the study. Patients will be identified from the National Veterans Affairs Health Care Network.
Sampling Method: Non-Probability Sample
Enrollment: 2313 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3431052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with metastatic castration-sensitive prostate cancer (mCSPC), who initiated Novel Hormonal Therapy (NHT) [abiraterone, apalutamide, or enzalutamide] in first line (1L) setting, any date (index date) from 01-Jan-2020 to 31-Dec-2022 were retrieved using the Veterans' Health Administration data for period of 01-Jan-2020 to 30-Sep-2023 (45 months). Retrospective data was evaluated from 22-Nov-2023 to 23-Apr-2024 (approximately 5 months) per objectives of the study.
Groups:
- Participant: NHT: Eligible participants who initiated NHT as therapy including 1L to treat mCSPC in real world setting from 01-January-2020 to 31-December-2022, their data were evaluated as per objectives of this study. No intervention was administered under this observational study.
Period: Overall Study
Arm/Group | Participant: NHT
Started | 2313
Completed | 2313
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included eligible participants whose data was retrieved and evaluated per objectives of this study.
Arm/Group | Participant: NHT
Number analyzed (Participants) | 2313
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-59 Years | 99
  Age: 60-69 Years | 451
  Age: 70-79 Years | 1206
  Age: Greater than or equal to (>=) 80 | 557
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2313
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data is reported as retrieved from medical records in accordance to protocol.
  Participants
    White, non-Hispanic | 1478
    Black | 522
    Hispanic | 114
    Other | 62
    Unknown | 137

OUTCOME MEASURES:

1. Primary Outcome: Duration of Therapy (DOT)
Description: DOT was defined as the time from the index date to the date of NHT discontinuation for any reason. Discontinuation of the current NHT was defined as a treatment gap of at least 90 days (the last day with days' supply before the gap as discontinuation date), the initiation of a new therapy, or death, whichever came first. Initiation of a new therapy was defined by switching to a different NHT, switching to or augmentation with different therapies. Participants who did not experience discontinuation were censored at the end of data availability. Index date was defined as the initiation date of NHT in 1L (any date) from 1-January-2020 to 31-December-2022. Retrospective data was retrieved using the Veterans' Health Administration data for period of 01-Jan-2020 to 30-Sep-2023 (45 months).
Time Frame: From start of index treatment to date of NHT discontinuation or censoring date, whichever came first, during maximum follow-up of 45 months
Population: Analysis population included eligible participants whose data was retrieved and evaluated per objectives of this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participant: NHT
Number analyzed (Participants) | 2313
Months | 18.5 [17.0 to 19.8]

2. Secondary Outcome: Time to Next Therapy (TTNT)
Description: TTNT was defined as the time from the index date to the initiation date of a new therapy. Initiation of a new therapy was defined by switching to a different NHT, switching to different therapies. Participants who did not initiate a new therapy were censored at the end of data availability or death, whichever came first. Index date was defined as the initiation date of NHT in 1L (any date) from 1-January-2020 to 31-December-2022. Retrospective data was retrieved using the Veterans' Health Administration data for period of 01-Jan-2020 to 30-Sep-2023 (45 months). Kaplan-Meier method was used for analysis.
Time Frame: From start of index treatment until date of new therapy, or censoring date, whichever came first; during maximum follow-up of 45 months
Population: Analysis population included eligible participants whose data was retrieved and evaluated per objectives of this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participant: NHT
Number analyzed (Participants) | 2313
Months | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient number of participants with event.

ADVERSE EVENTS:
Time Frame: Data for adverse events and death were not planned to be evaluated during the study; hence timeframe is not applicable
Description: Due to non-interventional nature of the study, minimum criteria for reporting an adverse event could not be met, hence adverse events were not planned to be evaluated. Thus, explaining 0 participant at risk.
Arm/Group | Participant: NHT
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT06151418/Prot_SAP_000.pdf